CLINICAL TRIAL: NCT00782626
Title: A Phase II Study of Everolimus (RAD001) for Children With Chemotherapy and/or Radiation-Refractory Progressive or Recurrent Low-Grade Gliomas
Brief Title: Everolimus (RAD001) for Children With Chemotherapy-Refractory Progressive or Recurrent Low-Grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); Pediatric Oncology Experimental Therapeutics Investigators' Consortium (Unknown)
Responsible Party: Principal Investigator, Karen D. Wright MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-001
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Glioma; Low-grade Glioma; Astrocytoma
Keywords: RAD001
MeSH Terms: conditions — Glioma; Astrocytoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- everolimus (Experimental): Patients rcvd oral everolimus 5.0 mg/m2/day for a 28-day treatment course up to a total of 12 courses (48 weeks) if a patient had stable disease except if toxicity was unacceptable. Two dose reductions were permitted (3.0 5.0 mg/m2/day and 2.0 mg/m2/day).
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus
  Other Names: RAD001

SUMMARY:
The purpose of this research study is to learn if the study drug RAD001 can shrink or slow the growth of low-grade gliomas. Additionally, the safety of RAD001 will be studied. RAD001 is a drug that may act directly on tumor cells by inhibiting tumor cell growth and proliferation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response of children with chemotherapy-refractory or progressive low-grade gliomas to everolimus. Secondary
* To evaluate pharmacogenetic polymorphisms of cytochrome P450 3A4 & 3A5 alleles and P-glycoprotein/MDR for their influence on the metabolism of everolimus in this patient population.
* To evaluate the role of Apolipoprotein E genotypes as predictors for development of hyperlipidemia during therapy with everolimus.
* To assess preliminary correlations of response with changes in pharmacodynamic parameters including p70s6 kinase activity in peripheral blood mononuclear cells.
* To describe the toxicity of everolimus when administered to this patient population.
* To characterize the pharmacokinetic profile of everolimus when administered to this patient population.

STATISTICAL DESIGN:

This study used a one-stage design to evaluate response to everolimus. If at least 3 responders are observed in 20 evaluable patients, then everolimus will be considered promising. If the true response rate is 5% (null hypothesis), the chance of concluding the treatment is active is 0.08 (Type I error). If the true response rate is 25% (alternative hypothesis), the chance of concluding the treatment is active is 0.91 (power).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic verification of one of the eligible diagnoses listed here: Astrocytoma variants; fibrillary, protoplasmic, mixed: Pilocytic astrocytoma; including pilomyxoid variants: Pleomorphic xanthoastrocytoma: infantile desmoplastic astrocytoma: ganglioglioma: oligodendroglial tumors: mixed glioma.
* Patients must have received at least one cancer-directed therapy and patients with allergies to carboplatin must have demonstrated progressive disease after cessation of therapy.
* Must have at least one measurable site of disease that has not been previously irradiated. If the patient has previous irradiation to the marker lesion(s), there must be evidence of progression since radiation treatment.
* Patients must be between 3 years of age and 21 years of age
* Karnofsky Performance Status of 50% or greater for patients less than 10 years of age or Lansky Score of 50% or greater for patients 10 and up.
* Participants must have recovered from the acute toxic effects of all prior chemotherapy or radiotherapy prior to entering the study. Refer to protocol for specific time restrictions with prior therapy completion.
* Adequate bone marrow function as defined in protocol
* Adequate renal function as defined in protocol
* Adequate liver function as defined in protocol
* Patients must have a fasting LDL cholesterol within the normal range per institutional guidelines
* Patients taking cholesterol lowering agent must be on a single medication and on a stable dose for at least 4 weeks
* Fasting serum cholesterol as outlined in protocol
* Patients must not be taking enzyme-inducing anticonvulsants
* Patients may not be currently receiving strong inhibitors of CYP3A4

Exclusion Criteria:

* Presence of NF1 by clinical examination or by genetic testing
* Patients who have had a major surgery or significant traumatic injury within 2 weeks of start of study drug, patients who have not recovered from teh side effects of any major surgery, or patients that may require major surgery during the course of the study
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled are allowed
* Evidence of plexiform neurofibroma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy
* Uncontrolled brain or leptomeningeal metastases from plexiform neurofibromas, malignant peripheral nerve sheath tumors, or other cancers (other than astrocytoma variants; fibrillary, protoplasmic, mixed: Pilocytic astrocytoma; including pilomyxoid variants: Pleomorphic xanthoastrocytoma: infantile desmoplastic astrocytoma: ganglioglioma: oligodendroglial tumors: mixed glioma), including patients who continue to require glucocorticoids for control of symptoms related to brain or leptomeningeal metastases.
* Other malignancies within the past three years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study (see protocol for examples)
* Known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Active, bleeding diathesis or oral anti-vitamin K medication (except low dose coumarin)
* Female patients who are pregnant or breast feeding
* Prior treatment with an mTOR inhibitor
* Known hypersensitivity to RAD001 or other rapamycins or to is excipients
* Dental braces or prosthesis that interferes with tumor imaging
* Patients with a positive history of Hepatitis B or Hepatitis C
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - Phoenix Children's Hospital Center for Cancer and Blood Disorders, Phoenix, Arizona
  - The Children's Hospital, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - John Hopkins Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New York University, New York, New York
  - Memorial Sloan-Kettering Cancer Institute, New York, New York
  - Doernbecher Children's Hospital Oregon Health & Science University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pts enrolled from 9 institutions over a two-year period (9/2009-9/2011).
Period: Overall Study
Arm/Group | Everolimus
Started | 23
Completed | 16
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 5
Not completed — Other Complicating Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants] — The analysis dataset is comprised of all eligible and treated patients.
  Participants
    <=18 years | 23
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 9 [3 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Overall response is classified as complete response (CR), partial response (PR), stable disease (SD) or Progressive Disease (PD) on therapy.Description: Overall response is classified as complete response (CR), partial response (PR), stable disease (SD) or Progressive Disease (PD) on therapy. Response for target lesions (up to5) is based on 3 dimensions with an elliptical model volume used: 0.5L*W*T; (L) tumor extent in plane perpendicular to the selected plane; (W) longest measurement of the tumor width; (T) transverse measurement perpendicular to the width. CR is disappearance all target and non-target lesions and no new lesions. PR is >/= 65% decrease in sum of the products (referent baseline). PD 40% or more increase in any target lesion (referent smallest product observed on therapy). SD is none of the above. PR and SD classification as long as absent new lesions and unequivocal progression for non-target lesions else PD.
Time Frame: Disease evaluations (MRI brain, including volumetric analysis) occurred at baseline, at the end of course 1, every 3 courses during treatment up to 12 courses and at early treatment discontinuation.
Population: The analysis dataset is comprised of all evaluable patients. All treated patients were evaluable.
Measure: Number; unit: participants
Arm/Group | Everolimus
Number analyzed (Participants) | 23
participants
  Partial Response | 2
  Stable Disease | 21

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Patients received up to 48 weeks of treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=23)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Infection-other (Infections and infestations) | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1
Neutrophils (Investigations) | 1
ALT, SGPT (Investigations) | 1
AST, SGOT (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=23)
Hemoglobin (Blood and lymphatic system disorders) | 6
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Middle ear, pain (Ear and labyrinth disorders) | 1
Hyopthyroidism (Endocrine disorders) | 1
Ocular-other (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Distention/bloating, abdominal (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 12
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 6
GI-other (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 2
Oral cavity, pain (Gastrointestinal disorders) | 2
Stomach, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Fever w/o neutropenia (General disorders) | 2
Pain-other (General disorders) | 2
Infection-other (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 9
Lymphopenia (Investigations) | 6
Neutrophils (Investigations) | 6
Platelets (Investigations) | 10
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (Investigations) | 3
AST, SGOT (Investigations) | 4
Hypercholesterolemia (Investigations) | 19
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Bicarbonate (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7
Hyperuricemia (Metabolism and nutrition disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No